CLINICAL TRIAL: NCT05987423
Title: A Phase III, Randomized, Double-Masked, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab in Participants With Moderate-to-Severe Thyroid Eye Disease
Brief Title: A Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab in Participants With Thyroid Eye Disease
Acronym: SatraGO-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP44467; 2023-503309-13-00 (EU CTIS Number)
Record Dates: First submitted 2023-07-05; First posted 2023-08-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease; TED
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — satralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Satralizumab (Experimental): In the Part I period, participants will receive satralizumab every 4 weeks (q4w) followed by proptosis response-based individualized treatment in Part II of the study
  Interventions: Drug: Satralizumab
- Placebo (Placebo Comparator): In the part I period, participants will receive placebo q4w followed by proptosis response-based individualized treatment in part II of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Satralizumab — Satralizumab will be administered by SC injection.
  Arms: Satralizumab
Drug: Placebo — Placebo will be administered by SC injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of subcutaneous (SC) satralizumab, a recombinant, humanized anti-interleukin-6 (IL-6) receptor monoclonal antibody, in participants with thyroid eye disease (TED).

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of TED based on CAS

Exclusion Criteria:

* Decrease in CAS or proptosis of >= 2 points or >= 2 mm, respectively, in the study eye between Screening and Study Baseline (Day 1)
* Requiring immediate surgical ophthalmological intervention or planning corrective surgery or irradiation during the course of the study, in the judgment of the investigator
* Identified pre-existing ophthalmic disease that, in the judgment of the investigator, would preclude study participation or complicate interpretation of study results, including corneal decompensation unresponsive to medical management and including ophthalmic diseases that will likely require prohibited therapy during the study
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes an individual's safe participation in and completion of the study
* Pregnant or breastfeeding, or intention of becoming pregnant during the study or within 3 months after the final dose of satralizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving ≥ 2mm Reduction in Proptosis from Baseline (Day 1) at Week 24 in the Study eye | Baseline, Week 24
  Provided there is no deterioration of proptosis [≥ 2 millimeters (mm) increase] in the fellow eye

SECONDARY OUTCOMES:
Change in Proptosis | Baseline, Week 24, Week 48 and from Week 24 to Week 48
Percentage of Participants Achieving ≥ 1 Grade Reduction/Improvement in Diplopia Among Participants with Baseline Diplopia | Baseline, Week 24, Week 48
Percentage of Participants Achieving Absence of Motility-induced Pain | Week 24
Percentage of Participants Achieving Absence of Spontaneous Pain | Week 24
Percentage of Participants with a ≥ 6 Point Improvement in the Visual Functioning and Appearance Sub-Scale Scores of the Graves Ophthalmopathy Quality of Life (GO-QoL) | Baseline, Week 24, Week 48 and from Week 24 to Week 48
  The GO-QoL is a 16-item self-administered questionnaire divided into two sub-scales and used to assess the perceived effects of TED by the participants on their: 1) Visual Functioning (questions 1-8); and 2) Appearance (questions 9-16). Both the subscales and overall score are transformed to a scale of 0 to 100. Higher total scores indicate better QoL.
Percentage of Participants Achieving Overall Response | Week 24. Week 48
Percentage of Participants Achieiving ≥2 Point Reduction in Clinical Activity Score (CAS) in the Study eye | Baseline, Week 24, Week 48
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to TED; 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active TED (ignore "equivocal" redness); 6. Chemosis; 7. Swelling of caruncle or plica. Each item is scored as 1 (present) or 0 (absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms). Higher scores indicate worse symptoms.
Percentage of Participants Acheiving CAS Value of 0 or 1 in the Study eye | Week 24
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to TED; 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active TED (ignore "equivocal" redness); 6. Chemosis; 7. Swelling of caruncle or plica. Each item is scored as 1 (present) or 0 (absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms). Higher scores indicate worse symptoms.
Percentage of Participants Achieving ≥ 10 point Improvement in Ocular Surface Disease Index (OSDI) Overall Scores | Baseline, Week 24
  The OSDI instrument is a validated dry eye questionnaire and consists of three main sections concerning ocular symptoms, visual function, and environmental factors. It comprises of 12 questions and for every question, participants selects a number between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time" with totals of score ranging from 0 to 100. Higher scores represents a worse disease index.
Change in OSDI Ocular Symptoms and Vision-related Function Subscale Scores | Baseline, Week 24
  The OSDI instrument is a validated dry eye questionnaire and consists of three main sections concerning ocular symptoms, visual function, and environmental factors. It comprises of 12 questions and for every question, participants selects a number between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time" with totals of score ranging from 0 to 100. Higher scores represents a worse disease index.
Change in Oxford Corneal Staining Scores | Baseline, Week 24
  Oxford corneal staining chart consists of a 6 point scale. Staining assessment will be based on the intensity of fluorescein staining, ranging from Grade 0 to V for each panel (Grade 0-I: normal; Grade II-III: mild to moderate; Grade IV-V: severe). Higher grade indicates worse worse disease index.
Percentage of Participants Achieving ≥ 2mm Reduction in Proptosis at Week 48 in the Study eye | Week 48
Percentage of Participants Requiring Surgical Intervention for TED | Up to Week 48
Percentage of Participants With Worsening of Proptosis by ≥ 2 mm | Baseline, Week 48 and from Week 24 to Week 48
Change in CAS | Baseline, Week 48 and from Week 24 to Week 48
  The CAS is a 7-item description of clinical activity, including: 1. Spontaneous orbital pain; 2. Gaze evoked orbital pain; 3. Eyelid swelling that is considered to be due to TED; 4. Eyelid erythema; 5. Conjunctival redness that is considered to be due to active TED (ignore "equivocal" redness); 6. Chemosis; 7. Swelling of caruncle or plica. Each item is scored as 1 (present) or 0 (absent) and scores for each item are summed for total score of 0 (no inflammatory symptoms) to 7 (most inflammatory symptoms). Higher scores indicate worse symptoms.
Percentage of Participants with Adverse Events (AEs), with Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5 (NCI CTCAE V5) | Baseline, Week 72
Serum Concentration of Satralizumab | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (46):
- United States (11):
  - Thrive Health Research LLC, Beverly Hills, California
  - UCSD Shiley Eye Center, La Jolla, California
  - Grene Vision Group, LLC, Wichita, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - 'Northwell Health Physician Partners Ophthalmology, Great Neck, New York
  - EyeHealth Northwest, Portland, Oregon
  - Austin Retina Associates, Austin, Texas
  - Eyelid Center of Utah, Salt Lake City, Utah
  - WVU Eye Institute, Morgantown, West Virginia
- Argentina (6):
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Centro Oftalmologico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Centrovision Mendoza, Mendoza
  - Grupo Laser Vision, Rosario
- Australia (3):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Centre For Eye Research Australia, East Melbourne, Victoria
- Medizinische Universitat Wien, Vienna, Austria
- Germany (6):
  - Charité-Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Augenheilkunde, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitatsklinikum Munster, Münster
  - Universitäts-Augenklinik Tübingen, Tübingen
- Hong Kong Eye Hospital, Mong Kok, Hong Kong
- Budapest Retina Associates Kft., Budapest, Hungary
- Italy (5):
  - A.O. U. Federico II, Napoli, Campania
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale Di Circolo E Fondazione Macchi, Varese, Lombardy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- Japan (10):
  - Aichi Medical University Hospital, Aichi
  - Kyushu University Hospital, Fukuoka
  - Social Medical Corporation Tenjinkai Shinkoga Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Kobe Kaisei Hospital Medical foundation, Hyōgo
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - University of Miyazaki Hospital, Miyazaki
  - Osaka Metropolitan University Hospital, Osaka
  - Olympia Eye Hospital, Tokyo
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore Eye Research Institute, Singapore

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Ezra D, Collins A, Haskova Z, Kuenzel T, Ida H, Triyatni M, Brittain C, Idowu O. Targeting IL-6 Receptor Signaling with Satralizumab in Thyroid Eye Disease: Design of the Phase 3 SatraGO-1 and SatraGO-2 Trials. Ophthalmol Ther. 2025 Dec;14(12):3119-3132. doi: 10.1007/s40123-025-01255-3. Epub 2025 Oct 9. PMID 41066062